CLINICAL TRIAL: NCT00885170
Title: A Phase IIa Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Effects of Odanacatib (MK-0822) on Bone Mineral Density (BMD) and Overall Safety in the Treatment of Osteoporosis in Postmenopausal Women Previously Treated With Alendronate
Brief Title: A Study to Evaluate the Safety, Tolerability, and Efficacy of Odanacatib (MK-0822) in Postmenopausal Women Previously Treated With a Bisphosphonate (MK-0822-042)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-042; 2009_578 (Other: Merck Registration Number); CTRI/2009/091/000218 (Registry Identifier: CTRI); 2008-008257-30 (EudraCT Number)
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — odanacatib; Cholecalciferol; Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Odanacatib 50 mg (Experimental): Odanacatib 50 mg tablets once weekly for 24 months. Vitamin D3 (dietary supplement), two 2800 IU tablets, taken once weekly for 24 months. Participants received calcium carbonate supplements as needed to ensure a daily calcium intake of 1200 mg.
  Interventions: Drug: Odanacatib; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium
- Placebo (Placebo Comparator): Placebo to odanacatib 50 mg tablets once weekly for 24 months. Vitamin D3 (dietary supplement), two 2800 IU tablets, taken once weekly for 24 months. Participants received calcium carbonate supplements as needed to ensure a daily calcium intake of 1200 mg.
  Interventions: Drug: Placebo; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium

INTERVENTIONS:
Drug: Odanacatib — Odanacatib 50 mg tablets once weekly for 24 months
  Arms: Odanacatib 50 mg
Drug: Placebo — Placebo to odanacatib 50 mg tablets once weekly for 24 months
  Arms: Placebo
Dietary Supplement: Vitamin D3 — Vitamin D3, two 2800 IU tablets, taken once weekly for 24 months
Dietary Supplement: Calcium — Participants will receive calcium carbonate supplements as needed to ensure a daily calcium intake of 1200 mg.

SUMMARY:
The study will evaluate the both the efficacy of odanacatib on Bone Mineral Density (BMD) and the safety of odanacatib for postmenopausal osteoporosis in patients previously treated with alendronate. The primary hypothesis of the trial is that treatment with odanacatib 50 mg once weekly will increase bone mineral density at the femoral neck compared to placebo at the end of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Has been postmenopausal for at least 5 years
* Has taken or is taking alendronate
* Agrees not to use medications for osteoporosis other than what is provided by the study

Exclusion Criteria:

* Has a history or evidence of hip fracture
* Has a history of cancer within 5 years of screening, except certain skin or cervical cancers.
* Has active parathyroid disease
* Has a history of thyroid disease not adequately controlled by medication
* Is taking anti-seizure medication and has abnormal calcium metabolism
* Has received any bisphosphonate other than alendronate for 20% of the last 3 years, or within 3 months of screening

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2009-04-13 (Actual); Primary Completion 2011-09-15 (Actual); Study Completion 2011-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Bonnick S, De Villiers T, Odio A, Palacios S, Chapurlat R, DaSilva C, Scott BB, Le Bailly De Tilleghem C, Leung AT, Gurner D. Effects of odanacatib on BMD and safety in the treatment of osteoporosis in postmenopausal women previously treated with alendronate: a randomized placebo-controlled trial. J Clin Endocrinol Metab. 2013 Dec;98(12):4727-35. doi: 10.1210/jc.2013-2020. Epub 2013 Sep 24. PMID 24064689

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated in 40 study centers located in the United States, Europe, South Africa, and Asia-Pacific.
Pre-assignment Details: Women ≥ 60 years of age who had been on, or were on, an alendronate therapy for postmenopausal osteoporosis were eligible to participate in this trial.
Groups:
- Odanacatib 50 mg: Odanacatib 50 mg tablets once weekly for 24 months. Vitamin D3 (dietary supplement), two 2800 IU tablets, taken once weekly for 24 months. Participants received calcium carbonate supplements as needed to ensure a daily calcium intake of approximately 1200 mg.
- Placebo: Placebo to odanacatib 50 mg tablets once weekly for 24 months. Vitamin D3 (dietary supplement), two 2800 IU tablets, taken once weekly for 24 months. Participants received calcium carbonate supplements as needed to ensure a daily calcium intake of approximately 1200 mg.
Period: Overall Study
Arm/Group | Odanacatib 50 mg | Placebo
Started | 124 | 122
Treated | 122 | 121
Completed | 86 | 99
Not Completed | 38 | 23
Not completed — Adverse Event | 12 | 4
Not completed — Excessive bone loss | 6 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 13 | 13

BASELINE CHARACTERISTICS:
Population: The baseline characteristics are displayed for the All-Participants-As-Treated Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Odanacatib 50 mg | Placebo | Total
Number analyzed (Participants) | 122 | 121 | 243
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.5 (6.7) | 71.1 (6.8) | 71.3 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 121 | 243
  Male | 0 | 0 | 0
Baseline DEXA Areal Bone Mineral Density T-score [Mean (Standard Deviation); unit: T-score] — Dual-energy X-ray absorptiometry (DEXA), Bone Mineral Density (BMD), T-score. T-Score is the difference between the BMD value and the average bone mass for sex-matched, healthy young adults; the difference being expressed in number of standard deviations; T-score based upon the normative database in use by the manufactures. A T-score of -1.0 or above is considered normal. More negative numbers are more indicative of osteoporosis.
  T-score
    Femoral Neck BMD T-score (122, 121, 243) | -2.35 (0.52) | -2.38 (0.48) | -2.36 (0.50)
    Hip Trochanter BMD T-score (122, 121, 243) | -1.91 (0.70) | -2.10 (0.79) | -2.00 (0.75)
    Total Hip BMD T-score (122, 121, 243) | -1.91 (0.62) | -2.05 (0.68) | -1.98 (0.65)
    Lumbar Spine BMD T-score (113, 116, 229) | -2.34 (1.10) | -2.49 (1.14) | -2.41 (1.12)
    1/3 Distal Forearm BMD T-score (114, 113, 227) | -2.62 (1.26) | -2.69 (1.10) | -2.65 (1.18)
Baseline Biochemical Markers of Bone Resorption and Bone Formation [Mean (Standard Deviation); unit: ng/mL]
  C-telopeptides of Type 1 collage (116, 117,233) | 0.19 (0.22) | 0.18 (0.14) | 0.19 (0.19)
  Serum bone specific alk. phosphatase (115,117,232) | 9.28 (4.63) | 9.41 (4.16) | 9.35 (4.39)
  Serum N-propeptide, T1 collagen (115, 117, 232) | 29.48 (28.18) | 27.79 (21.58) | 28.63 (25.03)
Urine N-Telopeptides/Creatinine Ratio [Mean (Standard Deviation); unit: nmol/mmol] — u-NTx/Cr (nmol/mmol), Odanacatib 50 mg N=115, Placebo N=114, Total N=229
  nmol/mmol | 26.00 (23.76) | 26.35 (18.08) | 26.17 (21.08)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Femoral Neck Bone Mineral Density (BMD) at Month 24
Description: BMD at the femoral neck was assessed by dual-energy X-ray absorptiometry (DXA) at baseline and Month 24.
Time Frame: Baseline and Month 24
Population: The population analyzed included all randomized, treated participants who had femoral neck BMD data at Baseline and Month 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 83 | 95
Percent Change | 1.73 [0.61 to 2.85] | -0.94 [-1.98 to 0.10]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; The primary hypothesis of the study was met if; in postmenopausal women previously treated with alendronate with low BMD, two years of treatment with odanacatib 50 mg significantly increased BMD at the femoral neck site compared to placebo (p-value < 0.001); Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; Difference in the Least Squares Means = 2.67, 95% CI 2-sided [1.17 to 4.17] — Baseline measurement and post-baseline percent changes from baseline, with fixed effects for treatment, time, duration of prior alendronate use (3-5 years, >5 years), geographic region, machine type (Lunar/Hologic) and treatment-by-time interaction

2. Primary Outcome: Percentage of Participants Experiencing One or More Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurred during the course of the study.
Time Frame: Up to 25 months
Population: The population analyzed included all participants who took at least one dose of study medication and were counted in the treatment group of the medication they actually took.
Measure: Number; unit: Percentage of participants
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 122 | 121
Percentage of participants | 68.0 | 73.6
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; Difference in Percentages vs. Placebo = -5.5, 95% CI 2-sided [-16.9 to 6.0] — Based on Miettinen & Nurminen method

3. Primary Outcome: Percentage of Participants Discontinuing Study Drug Due to an AE
Description: as for outcome 2
Time Frame: Up to 24 months
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 122 | 121
Percentage of participants | 9.0 | 3.3
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; Difference in the Percentage vs. Placebo = 5.7, 95% CI 2-sided [-0.4 to 12.6] — Based on Miettinen & Nurminen method

4. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD at Month 12
Description: BMD at the femoral neck was assessed by DXA at baseline and Month 12.
Time Frame: Baseline and 12 Months
Population: The population analyzed included all randomized, treated participants who had femoral neck BMD data at Baseline and Month 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 98 | 109
Percent Change | 0.60 [-0.32 to 1.53] | -0.28 [-1.16 to 0.59]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.166, Constrained longitudinal data analysis; Difference in the least Squares Means = 0.88, 95% CI 2-sided [-0.37 to 2.14] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percent Change From Baseline in Trochanter BMD at Month 24
Description: BMD at the trochanter was assessed by DXA at baseline and Month 24.
Time Frame: Baseline and 24 Months
Population: The population analyzed included all randomized, treated participants who had trochanter BMD data at Baseline and Month 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 83 | 95
Percent Change | 1.83 [0.34 to 3.32] | -1.35 [-2.73 to 0.03]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.002, Constrained longitudinal data analysis; Difference in the Least Squares Means = 3.18, 95% CI 2-sided [1.19 to 5.17] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percent Change From Baseline in Trochanter BMD at Month 12
Description: BMD at the trochanter was assessed by DXA at baseline and Month 12.
Time Frame: Baseline and 12 Months
Population: The population analyzed included all randomized, treated participants who had trochanter BMD data at Baseline and Month 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 98 | 109
Percent Change | 0.86 [-0.13 to 1.85] | -0.14 [-1.08 to 0.79]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.142, Constrained longitudinal data analysis; Difference in the Least Squares Means = 1.00, 95% CI 2-sided [-0.34 to 2.35] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Percent Change From Baseline in Total Hip BMD at Month 24
Description: BMD at the total hip was assessed by DXA at baseline and Month 24.
Time Frame: Baseline and 24 Months
Population: The population analyzed included all randomized, treated participants who had total hip BMD data at Baseline and Month 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 83 | 95
Percent Change | 0.83 [-0.13 to 1.80] | -1.87 [-2.77 to -0.97]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; Difference in the Least Squares Means = 2.70, 95% CI 2-sided [1.41 to 4.00] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Percent Change From Baseline in Total Hip BMD at Month 12
Description: BMD at the total hip was assessed by DXA at baseline and Month 12.
Time Frame: Baseline and 12 Months
Population: The population analyzed included all randomized, treated participants who had total hip BMD data at Baseline and Month 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 98 | 109
Percent Change | 0.26 [-0.41 to 0.94] | -0.80 [-1.44 to -0.16]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.023, cLDA; Difference in the Least Squares Means = 1.06, 95% CI 2-sided [0.15 to 1.98] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Month 24
Description: BMD at the lumbar spine was assessed by DXA at baseline and Month 24.
Time Frame: Baseline and 24 Months
Population: The population analyzed included all randomized, treated participants who had lumbar spine BMD data at Baseline and Month 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 80 | 89
Percent Change | 2.28 [1.30 to 3.25] | -0.30 [-1.21 to 0.62]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; Difference in the Least Squares Means = 2.57, 95% CI 2-sided [1.26 to 3.89] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Month 12
Description: BMD at the lumbar spine was assessed by DXA at baseline and Month 12.
Time Frame: Baseline and 12 Months
Population: The population analyzed included all randomized, treated participants who had lumbar spine BMD data at Baseline and Month 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 91 | 103
Percent Change | 0.69 [-0.03 to 1.40] | -0.12 [-0.79 to 0.56]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.103, cLDA; Difference in the Least Squares Means = 0.80, 95% CI 2-sided [-0.16 to 1.77] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Percent Change From Baseline in 1/3 Distal Forearm BMD at Month 24
Description: BMD at the 1/3 distal forearm was assessed by DXA at baseline and Month 24.
Time Frame: Baseline and 24 Months
Population: The population analyzed included all randomized, treated participants who had 1/3 distal forearm BMD data at Baseline and Month 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 80 | 86
Percent Change | -0.92 [-1.99 to 0.15] | -1.14 [-2.16 to -0.13]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.763, cLDA; Difference in the Least Squares Means = 0.22, 95% CI 2-sided [-1.23 to 1.67] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Percent Change From Baseline in 1/3 Distal Forearm BMD at Month 12
Description: BMD at the 1/3 distal forearm was assessed by DXA at baseline and Month 12.
Time Frame: Baseline and 12 Months
Population: The population analyzed included all randomized, treated participants who had 1/3 distal forearm BMD data at Baseline and Month 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 93 | 100
Percent Change | -0.11 [-1.11 to 0.89] | -0.49 [-1.44 to 0.47]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.578, cLDA; Difference in the Least Squares Means = 0.38, 95% CI 2-sided [-0.96 to 1.72] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Percent Change From Baseline in Log-Transformed Serum C-Telopeptides of Type I Collagen (s-CTx) at Month 24
Description: s-CTx is a biochemical marker of bone resorption.
Time Frame: Baseline and Month 24
Population: The population analyzed included all randomized, treated participants who had s-CTx data at Baseline and Month 24 but excluded participants due to important protocol deviations that may have substantially affected the results such as use of concomitant medication, lack of study medication compliance, and medical history.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 80 | 79
Percent change | 93.86 [69.42 to 121.82] | 83.70 [61.06 to 109.52]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.500, cLDA; Difference in the Least Squares Means = 10.16, 95% CI 2-sided [-19.39 to 39.72] — Log-transformed baseline and post-baseline measurements up to Month 24, with fixed effects for treatment, time, duration of prior alendronate use, geographical region, the interaction of time-by-treatment and the time-by-factor interactions

14. Secondary Outcome: Percent Change From Baseline in Log-Transformed s-CTx at Month 12
Description: s-CTx is a biochemical marker of bone resorption.
Time Frame: Baseline and Month 12
Population: The population analyzed included all randomized, treated participants who had s-CTx data at Baseline and Month 12 but excluded participants due to important protocol deviations that may have substantially affected the results such as use of concomitant medication, lack of study medication compliance, and medical history.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 91 | 100
Percent change | 62.27 [39.76 to 88.42] | 68.09 [45.58 to 94.08]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.709, cLDA; Difference in the Least Squares Means = -5.82, 95% CI 2-sided [-36.29 to 24.65] — [estimate comment as in outcome 13, analysis 1]

15. Secondary Outcome: Percent Change From Baseline in Log-Transformed Urine N-Telopeptides/Creatinine Ratio at Month 24
Description: N-Telopeptides of Type 1 Collagen to Urine Creatinine Ratio (u-NTx/Cr) is a biochemical marker of bone resorption.
Time Frame: Baseline and Month 24
Population: The population analyzed included all randomized, treated participants who had u-NTx/Cr data at Baseline and Month 24 but excluded participants due to important protocol deviations that may have substantially affected the results such as use of concomitant medication, lack of study medication compliance, and medical history.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 80 | 77
Percent change | -15.55 [-24.57 to -5.47] | 31.48 [17.60 to 47.01]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; Difference in the Least Squares Means = -47.04, 95% CI 2-sided [-62.40 to -31.67] — [estimate comment as in outcome 13, analysis 1]

16. Secondary Outcome: Percent Change From Baseline in Log-Transformed u-NTx/Cr at Month 12
Description: u-NTx/Cr is a biochemical marker of bone resorption.
Time Frame: Baseline and Month 12
Population: The population analyzed included all randomized, treated participants who had u-NTx/Cr data at Baseline and Month 12 but excluded participants due to important protocol deviations that may have substantially affected the results such as use of concomitant medication, lack of study medication compliance, and medical history.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 91 | 96
Percent change | -17.23 [-26.02 to -7.40] | 29.06 [15.94 to 43.66]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p < 0.001, cLDA; Difference in the Least Squares Means = -46.29, 95% CI 2-sided [-61.43 to -31.15] — [estimate comment as in outcome 13, analysis 1]

17. Secondary Outcome: Percent Change From Baseline in Log-Transformed Serum Bone-Specific Alkaline Phosphatase at Month 24
Description: Bone-Specific Alkaline Phosphatase (BSAP) is a biochemical marker of bone formation.
Time Frame: Baseline and Month 24
Population: The population analyzed included all randomized, treated participants who had BSAP data at Baseline and Month 24 but excluded participants due to important protocol deviations that may have substantially affected the results such as use of concomitant medication, lack of study medication compliance, and medical history.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 82 | 84
Percent change | 51.62 [39.49 to 64.79] | 40.65 [29.82 to 52.39]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.186, cLDA; Difference in the Least Squares Means = 10.96, 95% CI 2-sided [-5.29 to 27.22] — [estimate comment as in outcome 13, analysis 1]

18. Secondary Outcome: Percent Change From Baseline in Log-Transformed Serum BSAP at Month 12
Description: BSAP is a biochemical marker of bone formation.
Time Frame: Baseline and Month 12
Population: The population analyzed included all randomized, treated participants who had BSAP data at Baseline and Month 12 but excluded participants due to important protocol deviations that may have substantially affected the results such as use of concomitant medication, lack of study medication compliance, and medical history.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 94 | 101
Percent change | 30.91 [23.06 to 39.27] | 18.10 [11.29 to 25.32]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.015, cLDA; Difference in the Least Squares Means = 12.82, 95% CI 2-sided [2.54 to 23.10] — [estimate comment as in outcome 13, analysis 1]

19. Secondary Outcome: Percent Change From Baseline in Log-Transformed Serum N-Terminal Propeptide of Type I Collagen at Month 24
Description: Serum N-terminal propeptide of Type I collagen (s-P1NP) is a biochemical marker of bone formation.
Time Frame: Baseline and Month 24
Population: The population analyzed included all randomized, treated participants who had S-P1NP data at Baseline and Month 24 but excluded participants due to important protocol deviations that may have substantially affected the results such as use of concomitant medication, lack of study medication compliance, and medical history.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 82 | 85
Percent change | 90.70 [70.43 to 113.38] | 59.53 [43.10 to 77.84]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.011, cLDA; Difference in the Least Squares Means = 31.17, 95% CI 2-sided [7.13 to 55.21] — [estimate comment as in outcome 13, analysis 1]

20. Secondary Outcome: Percent Change From Baseline in Log-Transformed Serum N-terminal Propeptide of Type I Collagen at Month 12
Description: s-P1NP is a biochemical marker of bone formation.
Time Frame: Baseline and Month 12
Population: The population analyzed included all randomized, treated participants who had S-P1NP data at Baseline and Month 12 but excluded participants due to important protocol deviations that may have substantially affected the results such as use of concomitant medication, lack of study medication compliance, and medical history.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 94 | 101
Percent change | 80.37 [60.72 to 102.43] | 56.37 [39.86 to 74.82]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.059, cLDA; Difference in the Least Squares Means = 24.01, 95% CI 2-sided [-0.93 to 48.94] — [estimate comment as in outcome 13, analysis 1]

21. Secondary Outcome: Percent Change From Baseline in Log-Transformed Serum Calcium at Month 24
Description: Serum calcium is an index of calcium homeostasis.
Time Frame: Baseline and Month 24
Population: The population analyzed included all randomized, treated participants who had serum calcium data at Baseline and Month 24 but excluded participants due to important protocol deviations that may have substantially affected the results such as use of concomitant medication, lack of study medication compliance, and medical history.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 83 | 87
Percent Change | -2.40 [-3.23 to -1.56] | -2.51 [-3.31 to -1.70]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.846, cLDA; Difference in the Least Squares Means = 0.11, 95% CI 2-sided [-0.95 to 1.16] — [estimate comment as in outcome 13, analysis 1]

22. Secondary Outcome: Percent Change From Baseline in Log-Transformed Serum Phosphate at Month 24
Description: Serum phosphate is an index of mineral homeostasis.
Time Frame: Baseline and Month 24
Population: The population analyzed included all randomized, treated participants who had serum phosphate data at Baseline and Month 24 but excluded participants due to important protocol deviations that may have substantially affected the results such as use of concomitant medication, lack of study medication compliance, and medical history.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 83 | 86
Percent Change | 2.37 [-0.21 to 5.02] | 0.99 [-1.47 to 3.52]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.413, cLDA; Difference in the Least Squares Means = 1.38, 95% CI 2-sided [-1.91 to 4.67] — [estimate comment as in outcome 13, analysis 1]

23. Secondary Outcome: Percent Change From Baseline in Log-Transformed Serum Parathyroid Hormone at Month 24
Description: Serum parathyroid hormone (SPH) regulates calcium, phosphorus, and vitamin D levels in the blood.
Time Frame: Baseline and Month 24
Population: The population analyzed included all randomized, treated participants who had SPH data at Baseline and Month 24 but excluded participants due to important protocol deviations that may have substantially affected the results such as use of concomitant medication, lack of study medication compliance, and medical history.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 81 | 85
Percent Change | 4.38 [-4.08 to 13.58] | 10.28 [1.68 to 19.61]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.326, cLDA; Difference in the Least Squares Means = -5.91, 95% CI 2-sided [-17.66 to 5.85] — [estimate comment as in outcome 13, analysis 1]

24. Secondary Outcome: Percent Change From Baseline in Log-Transformed Serum 1,25 Dihydroxyvitamin D at Month 24
Description: 1,25 dihydroxyvitamin D [1,25(OH)2 D] is the active vitamin D metabolite and stimulates calcium absorption in the intestine.
Time Frame: Baseline and Month 24
Population: The population analyzed included all randomized, treated participants who had 1,25(OH)2 D data at Baseline and Month 24 but excluded participants due to important protocol deviations that may have substantially affected the results such as use of concomitant medication, lack of study medication compliance, and medical history.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 80 | 84
Percent Change | -5.23 [-15.32 to 6.05] | -6.71 [-16.25 to 3.93]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.835, cLDA; Difference in the Least Squares Means = 1.47, 95% CI 2-sided [-12.37 to 15.32] — [estimate comment as in outcome 13, analysis 1]

25. Secondary Outcome: Percent Change From Baseline in Log-Transformed Serum 25-Hydroxyvitamin D at Month 24
Description: The 25-hydroxy vitamin D [25(OH)D] test is the most accurate way to measure vitamin D. In the kidney, 25-hydroxy vitamin D is converted into 1,25 di-hydroxyvitamin D, the active vitamin D metabolite.
Time Frame: Baseline and Month 24
Population: The population analyzed included all randomized, treated participants who had 25(OH)D data at Baseline and Month 24 but excluded participants due to important protocol deviations that may have substantially affected the results such as use of concomitant medication, lack of study medication compliance, and medical history.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Odanacatib 50 mg | Placebo
Number analyzed (Participants) | 81 | 86
Percent Change | -2.57 [-8.16 to 3.37] | 0.57 [-5.01 to 6.47]
Statistical Analysis 1: Comparison: Odanacatib 50 mg vs Placebo; Test type: Superiority or Other; p = 0.376, cLDA; Difference in the Least Squares Means = -3.13, 95% CI 2-sided [-10.04 to 3.78] — [estimate comment as in outcome 13, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 25 months
Description: The APaT population included all participants who took at least one dose of study medication and were counted in the treatment group of the medication they actually took.
Arm/Group | Odanacatib 50 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 20/122 | 20/121
Other Adverse Events (participants affected / at risk) | 40/122 | 48/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Odanacatib 50 mg (N=122) | Placebo (N=121)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Pterygium (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster infection neurological (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Odanacatib 50 mg (N=122) | Placebo (N=121)
Bronchitis (Infections and infestations) | 7 (9) | 5 (5)
Nasopharyngitis (Infections and infestations) | 4 (4) | 8 (9)
Urinary tract infection (Infections and infestations) | 15 (18) | 20 (28)
Fall (Injury, poisoning and procedural complications) | 2 (4) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (13) | 14 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (15) | 13 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.